CLINICAL TRIAL: NCT00906932
Title: A Prospective Study Comparing the Trachview Videoscope to Standard Direct Laryngoscopy for Orotracheal Intubation
Brief Title: Comparison Study of a New Fiberoptic Intubation Device to Standard Intubation Techniques
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parker Medical (Unknown)
Responsible Party: Lynn P. Roppolo, Assistant Professor, University of Texas Southwestern
Other Study IDs: IRB# 022004-040
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: Fiberoptic intubation; direct laryngoscopy; Trachview; Comparison of a fiberoptic intubating videoscope to direct laryngoscopy.

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trachview videoscope, direct laryngoscopy: Each subject served as their own control - the Trachview videoscope and direct laryngoscopy was performed on by all subjects in a sequential fashion.
- See above: See above

SUMMARY:
This is a two part study comparing the Trachview videoscope to standard laryngoscopy in their ability to visualize the glottic opening. It is hypothesized that the glottic view is improved with the Trachview videoscope. Not only can the Trachview provide an alternative and often improved view of the airway, but can be used for teaching novice intubators. Furthermore, the Trachview requires minimal deviation from standard intubating techniques and thus, it is much easier to learn and use than many fiberoptic scopes currently available.

DETAILED DESCRIPTION:
This is a two part study. Part one: Adult airway mannequins were used. Subjects were medical students with no previous experience in intubation.

Part two: This was a convenience sample of patients undergoing elective surgery. All patients were consented. The subjects were physicians and nurse anesthetists who were going to be intubated in the operating room setting.

For both parts of the study, the subjects viewed the glottic opening using direct laryngoscopy followed or preceded by visualization of the glottic opening using the Trachview. The subjects were asked to score the amount of the glottic opening that could be visualized using the POGO (percent of glottic opening)score. Subjects were only given a very brief inservice on how to use the Trachview. Additional measurements such as presurgical airway assessments of the patients were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 years old and older

Exclusion Criteria:

* Individuals less than 18
* Pregnant patients
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students with no prior intubation experience and patients requiring intubation for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
In part one, the median POGO score for direct laryngoscopy was 25% and 90% for the TrachView™ (p<0.001). In part two, the POGO score for direct laryngoscopy was 100% in only 67 of the 122 cases while, for TrachView™ it was 100% in 109 (p<0.001). | 6 months

SECONDARY OUTCOMES:
In part one, the TrachView™ was "easy" to use by 68% of the trainees. In part two, the clinicians also reported that the TrachView™ was "easy" to use. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Kim HJ, Chung SP, Park IC, Cho J, Lee HS, Park YS. Comparison of the GlideScope video laryngoscope and Macintosh laryngoscope in simulated tracheal intubation scenarios. Emerg Med J. 2008 May;25(5):279-82. doi: 10.1136/emj.2007.052803. PMID 18434462
- [Result] Rowinsky EK, McGuire WP, Guarnieri T, Fisherman JS, Christian MC, Donehower RC. Cardiac disturbances during the administration of taxol. J Clin Oncol. 1991 Sep;9(9):1704-12. doi: 10.1200/JCO.1991.9.9.1704. PMID 1678781
- See also: This is the manufacturer of the Trachview videoscope — http://www.parkermedical.com